CLINICAL TRIAL: NCT06236295
Title: Investigating the Safety and Efficacy of SHR6508 Injection in the Treatment of Secondary Hyperparathyroidism in Hemodialysis Patients : A Multicenter, Long-term Clinical Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR6508-202
Record Dates: First submitted 2024-01-09; First posted 2024-02-01 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-01

CONDITIONS: Secondary Hyperparathyroidism (SHPT) in Subjects With Chronic Kidney Disease (CKD) on Hemodialysis
MeSH Terms: conditions — Hyperparathyroidism, Secondary

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR6508 (Experimental)
  Interventions: Drug: SHR6508

INTERVENTIONS:
Drug: SHR6508 — SHR6508 will be administered to all the eligible subjects

SUMMARY:
This is a multicenter, single-arm, long-term safety and tolerability trial. A total of 300 subjects with chronic kidney disease on hemodialysis are planned to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years of age or older
2. Subject understands the study procedures and agrees to participate in thestudy by giving written informed consent.
3. Subject must be receiving regular hemodialysis for at least 12 weeks
4. BMI ≥18 kg/m2 and ≤35 kg/m2
5. iPTH≥ 300pg/ mL

Exclusion Criteria:

1. Subject has received a a history of malignant tumor within 5 years prior to screening
2. Subject has a history of unstable angina, congestive heart failure (NYHA class III or IV), acute myocardial infarction, coronary angioplasty, or coronary arterial bypass grafting within the past 6 months prior to screening.
3. Postdialysis systolic blood pressure>180 mmHg and/or diastolic blood pressure>110 mmHg
4. Allergy to the investigational drug (SHR6508 injection) and any of its components or excipients
5. Subject has a history of drug use or excessive alcohol use within 6 months prior to screening
6. Female subjects who were pregnant or lactating
7. Other reasons for not participating as deemed by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of any adverse events that occurred during the clinical study | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Percent change from baseline in predialysis iPTH during the EAP | through study completion, an average of 1 year
Percent change from baseline in predialysis serum cCa during the EAP | through study completion, an average of 1 year
Percent change from baseline in predialysis serum phosphorus during the EAP | through study completion, an average of 1 year
Percent change from baseline in predialysis calcium-phosphorus product during the EAP | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided